CLINICAL TRIAL: NCT01225939
Title: A Randomised, Open-label, Three-way Cross-over, Phase I Study in Healthy Subjects to Assess the Pharmacokinetics of AZD8329 After Single Doses of the Oral Solid Formulation and the Oral Solution
Brief Title: A Study Conducted Over 3 Periods to Look at the Drug in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D2350C00007
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Healthy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 4-(4-(2-adamantylcarbamoyl)-5-tert-butyl-pyrazol-1-yl)benzoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Single Oral dose AZD8329 tablet (fasting)
  Interventions: Drug: AZD8329
- 2 (Experimental): Single Oral dose AZD8329 solution (fasting)
  Interventions: Drug: AZD8329
- 3 (Experimental): Single Oral dose AZD8329 tablet (Fed)
  Interventions: Drug: AZD8329

INTERVENTIONS:
Drug: AZD8329 — tablet
  Arms: 1; 3
Drug: AZD8329 — Solution
  Arms: 2

SUMMARY:
A study conducted over 3 periods to look at the drug in the body.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated written informed consent before any study specific procedures including consent for genetic research exploring genetic variations in CYP3A5
* suitable veins for cannulation or repeated venepuncture
* Subjects should have a body mass index (BMI) between 18 and 30 kg/m2

Exclusion Criteria:

* Abnormal vital signs (blood pressure and pulse) after 10 minutes supine rest, as judged by the investigator
* Prolonged QTcF >450 msec or shortened QTcF <350 msec or family history of long QT syndrome
* Suspicion of known Gilbert's disease
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Compare the pharmacokinetics (Cmax and AUC) of the oral solution and the oral solid formulation of AZD8329. | Information will be collected during 48h after each dose.

SECONDARY OUTCOMES:
Explore the effect of food on the pharmacokinetics (Tmax, T1/2 and CL/F) of AZD8329 oral solid formulation. | Information will be collected during 48h after dose.
Investigate the safety and tolerability of AZD8329 administered as two different oral formulations.(Safety variables: Adverse events, Vital Signs, Clinical chemistry, Electrocardiogram (p ECG)) | Adverse event will be collected from first dose to last visit . Clinical chemistry, Vital Signs and pECG's will be collected at all 5 visits

CONTACTS AND LOCATIONS:
Overall Officials: J Ritter, BM BCh, MRCP, FRCP, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital; Dr. Mirjana Kujacic, Study Chair — AstraZeneca Mölndal; Jan Eriksson, MD PhD, Study Director — AstraZeneca Sweden
Locations (1):
- Research Site, London Bridge, United Kingdom